CLINICAL TRIAL: NCT05289128
Title: Predicting Outcomes From HD-tDCS Intervention in Long COVID-19 Using Electroencephalographic Biomarkers and Machine Learning Approach.
Brief Title: EEG as Predictor of HD-tDCS Effectiveness in Long COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, Principal Investigator, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LongCOVID/EEG/HDtDCS
Record Dates: First submitted 2022-03-16; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Coronavirus COVID-19; Respiratory Infection
Keywords: Transcranial direct current stimulation; Non-invasive brain stimulation; Electroencephalography; Machine Learning; COVID-19 Respiratory Infection; Long COVID
MeSH Terms: conditions — Respiratory Tract Infections; Post-Acute COVID-19 Syndrome | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group/ Active HD-tDCS (Experimental): Patients randomly enrolled in this group will receive 10 sessions of anodal HD-tDCS stimulation on cortical representation zone of left diaphragmatic motor cortex associated to respiratory training; for 20 minutes (each session) with a 2mA intensity. The electrical current will be delivered with a ramp-up time of 30 s, held at 3mA for 20 min, and then ramped down over 30 s.
  Interventions: Device: Experimental group
- Control Group / Sham Group (Sham Comparator): Patients enrolled in this group condition will receive 10 sessions of anodal stimulation on cortical representation zone of left diaphragmatic motor cortex using HD-tDCS associated to respiratory training; for 20 minutes (each session) with a 2mA intensity. In the sham condition, the device will provide a 30-second ramp-up followed immediately by a 30-second ramp down.
  Interventions: Device: Sham Control

INTERVENTIONS:
Device: Experimental group — 10-sessions of anodal HD-tDCS ( tDCS 1x1, developed by Soterix Medical Inc.) associated to respiratory training; for 20 minutes (each session). It will be delivered a 3mA intensity electrical current accordingly 10/20 International System on cortical representation zone of left diaphragmatic motor cortex using HD-tDCS.
  Other Names: Active HD-tDCS
  Arms: Experimental Group/ Active HD-tDCS
Device: Sham Control — 10-sessions of anodal HD-tDCS( tDCS 1x1, developed by Soterix Medical Inc.) associated to respiratory training; for 20 minutes (each session) with a 3mA intensity.The device will provide a 30-second ramp-up followed immediately by a 30-second ramp down.
  Other Names: Control Group
  Arms: Control Group / Sham Group

SUMMARY:
COVID-19 is an infectious disease which presents a heterogenous clinical presentation. Recent investigations suggest that people who were infected by COVID-19 often develop physical disabilities (i.e. pain, fatigue) and neurological complications after hospital discharge. Many therapeutic approaches such as transcranial direct current stimulation (tDCS) have been proposed to minimize functional and structural impairments. Electroencephalogram (EEG) has been used in this population to assess electrophysiological changes in the brain. However, evidences about EEG utilization as efficacy predictor of tDCS in COVID-19 people rest inconclusive.Our objective is to evaluate EEG as neurobiological predictor marker of tDCS efficacy on fatigue, pain, quality of life, self-efficacy and functional capacity in the chronic phase of COVID-19.

DETAILED DESCRIPTION:
A double-blinded randomized clinical trial will be carried to analyse the EEG as neurobiological predictor marker of HD-tDCS 4x1 in patients in long COVID-19. This study is in accordance with the CONSORT guidelines, which will investigate the effectiveness of treatment with HD-tDCS.

Patients who had a medical diagnosis of COVID-19, clinically stable, able to respond to simple commands, able to walk for six minutes and who sign study consent form will be enrolled. Those who present associated neurological diseases, pregnant, users of psychoactive drugs, patients who have metallic implants, electronic devices, pacemakers, or epileptic patients will be excluded.

Patients will be allocated randomly to the experimental group or sham control. Sessions for experimental group consist of anodal HD-tDCS on Left diaphragmatic primary motor cortex associated to respiratory training (10 sessions, 3mA, 20 minutes/session). In the sham condition, the device provided a 30-second ramp-up period to the full 3 mA, followed immediately by a 30-second ramp down.

Patients will be assessed in three moments: pre-treatment, post-treatment and after 30 days treatment ending (follow-up).

ELIGIBILITY:
Patients who had a medical diagnosis of COVID-19, clinically stable, able to respond to simple commands, able to walk for six minutes and who sign study consent form will be enrolled. Those who present associated neurological diseases, pregnant, users of psychoactive drugs, patients who have metallic implants, electronic devices, pacemakers, or epileptic patients will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-06-25 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Responders and non-responders to treatment with HD-tDCS | From date of randomization up to 5 weeks
  Identification of responders and non-responders according to the scores fatigue measured using MFIS-BR.

SECONDARY OUTCOMES:
Neurophysiological characteristics and biomarkers recorded by EEG | Assessed one week before intervention beginning (T0);
  The EEG data will be retrospectively examined by comparing the two groups (responders and non-responders), identifying possible neurophysiological characteristics and biomarkers related to frequency bands and connectivity that could be characterized as possible markers of response to treatment, predicting which ones are most likely to respond.
Pain Level | From date of randomization (1 week before intervention beginning ) up to 5 weeks (T1) and up to 10 weeks (T2; follow-up)
  Pain level will be evaluated through McGill questionnaire considering pain multifactorial characteristics.
Functional Capacity | From date of randomization (1 week before intervention beginning ) up to 5 weeks (T1) and up to 10 weeks (T2; follow-up)
  Functional capacity will be evaluated by Lawton and Brody scale and also by 6 minutes walking test.
Quality of Life | From date of randomization (1 week before intervention beginning ) up to 5 weeks (T1) and up to 10 weeks (T2; follow-up)
  Quality of life will be measured through Brazilian version of World Health Organization Quality of Life.
Pulmonary Function | From date of randomization (1 week before intervention beginning ) up to 5 weeks (T1) and up to 10 weeks (T2; follow-up)
  This outcome will be assessed through spirometry, assessment of maximal inspiratory pressure and respiratory endurance.
Body Composition | From date of randomization (1 week before intervention beginning ) up to 5 weeks (T1) and up to 10 weeks (T2; follow-up)
  Body composition analysis will be carried out by bioelectrical impedance analysis.
Anxiety | From date of randomization (1 week before intervention beginning ) up to 5 weeks (T1) and up to 10 weeks (T2; follow-up)
  Anxiety level will be evaluate through Hamilton Anxiety Rating Scale which measures the severity of anxiety symptoms.
Depression | From date of randomization (1 week before intervention beginning ) up to 5 weeks (T1) and up to 10 weeks (T2; follow-up)
  Depression will be assessed by Beck's Depression Inventory.
Self-efficacy | From date of randomization (1 week before intervention begining) up to 5 weeks (T1)
  Self-efficacy will be evalluated through the Self-efficacy manage chronic disease 6-item scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Paraíba,Department of Psychology, João Pessoa, Paraíba, Brazil